CLINICAL TRIAL: NCT06769204
Title: Safety and Efficacy of Lidocaine Prilocaine Spray in Reducing Pain During Hysterosalpingography in Women With Primary Infertility
Brief Title: Lidocaine Prilocaine Spray in Reducing Pain During Hysterosalpingography in Women With Primary Infertility
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP SPRAY HSG
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine prilocaine (Experimental)
  Interventions: Drug: EMLA SPRAY
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMLA SPRAY — 2 puffs of lidocaine-prilocaine spray into the cervix and cervical canal 5 minutes before the procedure
  Other Names: 2 puffs into
  Arms: lidocaine prilocaine
Drug: Placebo — 2 puffs of saline into the cervix and cervical canal 5 minutes before the procedure
  Arms: placebo

SUMMARY:
We aim to assess the Safety and Efficacy of Cervical Lidocaine Prilocaine Spray in Reducing Pain During Hysterosalpingography in women with primary infertility

DETAILED DESCRIPTION:
We aim to assess the Safety and Efficacy of Cervical Lidocaine Prilocaine Spray in Reducing Pain During Hysterosalpingography in Women with Primary Infertility.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years. Diagnosed with primary infertility (no prior pregnancy after at least 12 months of unprotected intercourse) and scheduled for HSG as part of infertility evaluation.

Exclusion Criteria:

* Known allergy or hypersensitivity to lidocaine, prilocaine, or any components of the spray.
* Current pregnancy or suspicion of pregnancy.
* Active pelvic inflammatory disease or history of severe pelvic infections within the last 6 months.
* Use of systemic analgesics, sedatives, or anesthetics within 24 hours prior to the procedure.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
pain during Cervical instrumentation of the tenaculum and cannula | 1 minute
  pain is measured using 10 cm VISUAL Analog scale where 0 denotes no pain and 10 maximum pain felt

SECONDARY OUTCOMES:
pain At the end of uterine filling | 5 minutes
  pain is measured using 10 cm VISUAL Analog scale where 0 denotes no pain and 10 maximum pain felt

IPD SHARING:
Plan to Share IPD: Undecided